CLINICAL TRIAL: NCT00169845
Title: Beta-carotene and Alpha-tocopherol Chemoprevention of Second Primary Malignancies in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Cancer Trials Group (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Isabelle Bairati, Professor (MD, PhD), Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 27370; NCIC-4738 (Other Grant/Funding Number: National Cancer Institute of Canada); NCIC-8176 (Other Grant/Funding Number: National Cancer Institute of Canada); NCIC-13211 (Other Grant/Funding Number: National Cancer Institute of Canada); NCIC-019502 (Other Grant/Funding Number: National Cancer Institute of Canada); 1R03CA141615-01 (NIH); 018100 (Other Grant/Funding Number: National Cancer Institute of Canada)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Neoplasms
Keywords: chemoprevention trial; antioxidant; alpha-tocopherol; beta-carotene; second primary cancer; head and neck cancer; adverse effect of radiation therapy; quality of life; mortality; cancer free survival; cancer recurrence
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; Head and Neck Neoplasms; Radiation Injuries | interventions — alpha-Tocopherol; beta Carotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alpha-Tocopherol and Beta-Carotene (Experimental): Patients received a daily supplementation of alpha-tocopherol (one capsule of 400 IU dl-alpha-tocopherol) and beta-carotene (one capsule of 30 mg) for 3 years after the end of radiation therapy. Due to ethical concerns, the beta-carotene supplementation was stopped during the trial (after the randomization of 156 patients). See details in JNCI, 2005: 97 (7), 481-8.
  Interventions: Dietary Supplement: Alpha-Tocopherol and Beta-Carotene
- Placebo (Placebo Comparator): Patients received two capsules of placebos per day during 3 years. When the beta-carotene was stopped, they received only one capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha-Tocopherol and Beta-Carotene — Provided by Roche Vitamins Inc.
  Arms: Alpha-Tocopherol and Beta-Carotene
Dietary Supplement: Placebo — Provided by Roche Vitamins Inc
  Arms: Placebo

SUMMARY:
Epidemiologic studies suggest that low dietary intakes and low plasma concentrations of antioxidant vitamins and minerals are associated with increased risks of cancer, especially for epidermoid tumors. Patients with stage I or II head and neck cancer have a good prognosis, with a 5-year relative survival of 60% to 90%, depending of the tumor site. However, the benefit of treatment is often compromised by the occurrence of second primary cancers, which develop in 20% of patients during the first 5 years after diagnosis. We conducted a randomized chemoprevention trial among patients with head and neck cancer treated by radiation therapy to determine whether supplementation combining two antioxidants, alpha-tocopherol and beta-carotene, could reduce the incidence of second primary cancers in this patient population (primary objective of the trial). This study was conducted with funds from the NCIC (#008176,004738,013211) and was completed.

In this cohort of head and neck cancer patients, we evaluated whether nine potential prognostic serum markers measured at the time of diagnosis were related to recurrence, occurence of second primary cancers and survival. This study was conducted with funds from the NCIC (#018100) and was completed.

Presently, we evaluate genetic polymorphisms(GWAS) associated with prognosis (NCIC grant #019502). We also assess the relationship between vitamin D (dietary intake, serum level, and genetic polymorphisms of key vitamin D-related genes) and head and neck long-term outcomes (NCI grant #1R03CA141615-01).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented stage I or II head and neck cancer

Exclusion Criteria:

* Karnofsky performance score of less than 60
* Multiple primary head and neck cancer
* History of cancer
* Severe cardiovascular disease
* Inadequate renal, hepatic or hematologic function
* Anticoagulant therapy
* Pregnancy
* Average daily supplement intake of beta-carotene or vitamin E in the preceding year greater than 6.0 mg and 50 IU, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 1994-10; Primary Completion 2003-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Second primary cancers | Immediately and 1 month after radiation therapy, every 6 months during the 3 years following the end of radiation therapy, and then once a year until June 30, 2003

SECONDARY OUTCOMES:
Acute and late side-effects of radiation therapy | During radiation therapy (RT), at the end of RT, one month after RT, six months after RT and 1 year after RT
Quality of life | Baseline, at the end of radiation therapy (RT), 1, 6,12,24 and 36 months after RT
Recurrence | Immediately and 1 month after radiation therapy, every 6 months during the 3 years following the end of radiation therapy, and then once a year until June 30, 2003
Cancer free survival | Immediately and 1 month after radiation therapy, every 6 months during the 3 years following the end of radiation therapy, and then once a year until June 30, 2003
  Without recurrence and without second primary cancer
Overall survival | Every year
Disease free survival | Immediately and 1 month after radiation therapy, every 6 months during the 3 years following the end of radiation therapy, and then once a year until June 30, 2003
  Alive and without recurrence
Survival until death from first cancer | every year
Survival until death from second primary cancer | Every year
Survival until death from non-cancer causes | Every year

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Bairati, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University Cancer Research Center, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
A letter was sent to each participant.

REFERENCES:
- [Result] Bairati I, Meyer F, Gelinas M, Fortin A, Nabid A, Brochet F, Mercier JP, Tetu B, Harel F, Abdous B, Vigneault E, Vass S, Del Vecchio P, Roy J. Randomized trial of antioxidant vitamins to prevent acute adverse effects of radiation therapy in head and neck cancer patients. J Clin Oncol. 2005 Aug 20;23(24):5805-13. doi: 10.1200/JCO.2005.05.514. Epub 2005 Jul 18. PMID 16027437
- [Result] Bairati I, Meyer F, Gelinas M, Fortin A, Nabid A, Brochet F, Mercier JP, Tetu B, Harel F, Masse B, Vigneault E, Vass S, del Vecchio P, Roy J. A randomized trial of antioxidant vitamins to prevent second primary cancers in head and neck cancer patients. J Natl Cancer Inst. 2005 Apr 6;97(7):481-8. doi: 10.1093/jnci/dji095. PMID 15812073
- [Result] Bairati I, Meyer F, Jobin E, Gelinas M, Fortin A, Nabid A, Brochet F, Tetu B. Antioxidant vitamins supplementation and mortality: a randomized trial in head and neck cancer patients. Int J Cancer. 2006 Nov 1;119(9):2221-4. doi: 10.1002/ijc.22042. PMID 16841333
- [Result] Meyer F, Bairati I, Jobin E, Gelinas M, Fortin A, Nabid A, Tetu B. Acute adverse effects of radiation therapy and local recurrence in relation to dietary and plasma beta carotene and alpha tocopherol in head and neck cancer patients. Nutr Cancer. 2007;59(1):29-35. doi: 10.1080/01635580701397590. PMID 17927499
- [Result] Sackett MK, Bairati I, Meyer F, Jobin E, Lussier S, Fortin A, Gelinas M, Nabid A, Brochet F, Tetu B. Prognostic significance of cyclooxygenase-2 overexpression in glottic cancer. Clin Cancer Res. 2008 Jan 1;14(1):67-73. doi: 10.1158/1078-0432.CCR-07-2028. PMID 18172254
- [Result] Meyer F, Fortin A, Gelinas M, Nabid A, Brochet F, Tetu B, Bairati I. Health-related quality of life as a survival predictor for patients with localized head and neck cancer treated with radiation therapy. J Clin Oncol. 2009 Jun 20;27(18):2970-6. doi: 10.1200/JCO.2008.20.0295. Epub 2009 May 18. PMID 19451440
- [Result] Meyer F, Samson E, Douville P, Duchesne T, Liu G, Bairati I. Serum prognostic markers in head and neck cancer. Clin Cancer Res. 2010 Feb 1;16(3):1008-15. doi: 10.1158/1078-0432.CCR-09-2014. Epub 2010 Jan 26. PMID 20103685
- [Result] Nourissat A, Bairati I, Samson E, Fortin A, Gelinas M, Nabid A, Brochet F, Tetu B, Meyer F. Predictors of weight loss during radiotherapy in patients with stage I or II head and neck cancer. Cancer. 2010 May 1;116(9):2275-83. doi: 10.1002/cncr.25041. PMID 20187097
- [Result] Meyer F, Liu G, Douville P, Samson E, Xu W, Adjei A, Bairati I. Dietary vitamin D intake and serum 25-hydroxyvitamin D level in relation to disease outcomes in head and neck cancer patients. Int J Cancer. 2011 Apr 1;128(7):1741-6. doi: 10.1002/ijc.25496. Epub 2010 Jun 7. PMID 20533282
- [Result] Meyer F, Bairati I, Fortin A, Gelinas M, Nabid A, Brochet F, Tetu B. Interaction between antioxidant vitamin supplementation and cigarette smoking during radiation therapy in relation to long-term effects on recurrence and mortality: a randomized trial among head and neck cancer patients. Int J Cancer. 2008 Apr 1;122(7):1679-83. doi: 10.1002/ijc.23200. PMID 18059031
- [Result] Nourissat A, Bairati I, Fortin A, Gelinas M, Nabid A, Brochet F, Tetu B, Meyer F. Factors associated with weight loss during radiotherapy in patients with stage I or II head and neck cancer. Support Care Cancer. 2012 Mar;20(3):591-9. doi: 10.1007/s00520-011-1132-x. Epub 2011 Mar 20. PMID 21424341
- [Result] Meyer F, Fortin A, Wang CS, Liu G, Bairati I. Predictors of severe acute and late toxicities in patients with localized head-and-neck cancer treated with radiation therapy. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1454-62. doi: 10.1016/j.ijrobp.2011.04.022. Epub 2011 Jun 2. PMID 21640495
- [Result] Azad AK, Bairati I, Samson E, Cheng D, Cheng L, Mirshams M, Savas S, Waldron J, Wang C, Goldstein D, Xu W, Meyer F, Liu G. Genetic sequence variants and the development of secondary primary cancers in patients with head and neck cancers. Cancer. 2012 Mar 15;118(6):1554-65. doi: 10.1002/cncr.26446. Epub 2011 Aug 25. PMID 22009713
- [Result] Azad AK, Bairati I, Samson E, Cheng D, Mirshams M, Qiu X, Savas S, Waldron J, Wang C, Goldstein D, Xu W, Meyer F, Liu G. Validation of genetic sequence variants as prognostic factors in early-stage head and neck squamous cell cancer survival. Clin Cancer Res. 2012 Jan 1;18(1):196-206. doi: 10.1158/1078-0432.CCR-11-1759. Epub 2011 Nov 10. PMID 22076708
- [Result] Azad AK, Bairati I, Qiu X, Huang H, Cheng D, Liu G, Meyer F, Adjei A, Xu W. Genetic sequence variants in vitamin D metabolism pathway genes, serum vitamin D level and outcome in head and neck cancer patients. Int J Cancer. 2013 Jun 1;132(11):2520-7. doi: 10.1002/ijc.27946. Epub 2012 Dec 14. PMID 23169318
- [Result] Azad AK, Bairati I, Qiu X, Girgis H, Cheng L, Waggott D, Cheng D, Mirshams M, Ho J, Fortin A, Vigneault E, Huang SH, O'Sullivan B, Waldron J, Boutros PC, Goldstein D, Meyer F, Xu W, Liu G. A genome-wide association study of non-HPV-related head and neck squamous cell carcinoma identifies prognostic genetic sequence variants in the MAP-kinase and hormone pathways. Cancer Epidemiol. 2016 Jun;42:173-80. doi: 10.1016/j.canep.2016.05.001. Epub 2016 May 9. PMID 27173062